CLINICAL TRIAL: NCT06962189
Title: The Efficacy and Safety of Sintilimab Plus Chemotherapy in Surgical Conversion for Patients With Unresectable Stage IIIB-IIIC NSCLC: A Prospective, Single-Arm, Phase II Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITRAD
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer (Stage III)
Keywords: NSCLC; IIIB-IIIC stage; conversion therapy; chemoimmunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemoimmunotherapy induction group (Experimental): For treatment-naive patients with unresectable IIIB-IIIC stage NSCLC, 3-4 cycles of induction chemoimmunotherapy, then radical pulmonary resection± definitive radiotherapy for metastatic lymph nodes, then PD-1 inhibitor maintenance therapy for 1 year
  Interventions: Drug: chemoimmunothrapy

INTERVENTIONS:
Drug: chemoimmunothrapy — Patients will receive 3-4 cycles of induction therapy with Sintilimab combined with platinum-based doublet chemotherapy, followed by multidisciplinary team (MDT) evaluation. For patients deemed eligible for radical lung primary lesion resection, surgery should be performed within 4-6 weeks after completing the final cycle of chemoimmunotherapy. The timing of radiotherapy for metastatic lymph nodes will be determined by MDT discussion. If deemed inoperable after induction therapy by MDT, definitive radiotherapy will be administered subsequently. All patients, in the absence of contraindications, will receive PD-1 inhibitor maintenance therapy for 1 year following local treatment.

SUMMARY:
This study aimed to evaluate the conversion rate to curative-intent treatment in patients with unresectable stage IIIB-IIIC non-small cell lung cancer (NSCLC) following induction therapy with PD-1 blockade combined with chemotherapy, and to assess progression-free survival (PFS) in these patients who underwent curative-intent treatment .

DETAILED DESCRIPTION:
This study is a prospective phase II trial designed to evaluate the safety and efficacy of radical resection of the primary lung lesion combined with radical radiotherapy for metastatic lymph nodes, followed by sequential PD-1 inhibitor consolidation therapy, in treatment-naïve patients with unresectable stage IIIB-IIIC non-small cell lung cancer (NSCLC) who received induction therapy with Sintilimab plus platinum-based doublet chemotherapy. The study plans to enroll 39 pathologically confirmed, driver mutation-negative, treatment-naïve stage IIIB-IIIC NSCLC patients. Eligible patients will receive 3-4 cycles of Sintilimab combined with platinum-based doublet induction chemotherapy, followed by assessment for feasibility of radical lung resection.The primary objectives are to evaluate: (1)The conversion rate to curative-intent treatment (radical resection and/or definitive radiotherapy) after induction chemoimmunotherapy in treatment-naïve unresectable stage IIIB-IIIC NSCLC patients; (2) Progression-free survival (PFS) in patients who undergo curative-intent treatment post-induction. Secondary objectives include observation of adverse event rates, objective response rate (ORR), major pathological response (MPR), PFS, overall survival (OS), and exploration of biomarkers associated with treatment efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients voluntarily participate in this study and sign informed consent forms (including consent for relevant testing of collected biological samples).

  2. Histologically or cytologically confirmed NSCLC with no prior antitumor therapy (including systemic medications or local treatments).

  3.Treatment-naïve patients with unresectable stage IIIB-IIIC NSCLC. 4. Evaluated by a multidisciplinary team (MDT): Surgical resection is not the current preferred treatment option, but radical resection of the primary lung lesion is feasible after induction chemoimmunotherapy, and metastatic contralateral/supraclavicular lymph nodes (if present) are amenable to definitive radiotherapy.

  5. Aged 18-75 years, regardless of gender. 6. ECOG performance status 0-1. 7. At least one measurable lesion per RECIST v1.1 criteria. 8. All suspicious mediastinal lymph nodes (e.g., pathologically enlarged or PET-CT-suggested malignancy) must undergo pathological confirmation via endobronchial ultrasound (EBUS), thoracoscopy, or mediastinoscopy if technically feasible.

  9. Pulmonary function (e.g., FVC, FEV1, TLC, FRC, DLco) deemed adequate for planned lung resection by MDT assessment.

  10. Absence of comorbidities that would elevate surgical risk to unacceptable levels.

  11. Adequate organ function within 14 days prior to enrollment (no blood components, growth factors, or corrective therapies allowed during this period): Absolute neutrophil count ≥1.5×10⁹/L, Platelets ≥100×10⁹/L, Hemoglobin ≥90 g/L, Serum albumin ≥35 g/L TSH ≤1×ULN, Total bilirubin ≤1.5×ULN, ALT/AST ≤3×ULN, INR ≤1.5 or PT ≤1.5×ULN, Serum creatinine ≤1.5×ULN 12. Non-sterilized or premenopausal female patients must use contraception (e.g., IUD, oral contraceptives, condoms) during the study and for 3 months post-treatment. Non-sterilized females must have a negative serum/urine HCG test within 72 hours before enrollment, be non-lactating, and male patients with fertile partners must use effective contraception during the trial and for 3 months after the last dose.

Exclusion Criteria:

* 1. Patients with NSCLC harboring driver mutations (e.g., EGFR, ALK, ROS1). 2. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 therapies targeting T-cell co-stimulatory pathways.

  3. History of concurrent or other malignancies within the past 3 years (except cured basal cell carcinoma of the skin or cervical carcinoma in situ).

  4. Active hepatitis B/C with poor response to antiviral therapy. 5. Active autoimmune diseases or history of autoimmune disorders (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism; vitiligo is permitted; childhood asthma resolved without intervention in adulthood is allowed; asthma requiring bronchodilators is excluded).

  6. Current use of immunosuppressants or systemic corticosteroids (>10 mg/day prednisone equivalent) for immunosuppression within 2 weeks prior to enrollment.

  7. Poorly controlled hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg) or uncontrolled cardiac conditions: NYHA class ≥II heart failure, Unstable angina, Myocardial infarction within 1 year, Clinically significant supraventricular/ventricular arrhythmias requiring treatment, QTc >450 ms (men) or >470 ms (women).

  8.Coagulopathy (INR >2.0, PT >16 s), bleeding tendency, or ongoing thrombolytic/anticoagulant therapy (prophylactic low-dose aspirin or LMWH is permitted).

  9.Arterial/venous thrombotic events within 6 months (e.g., cerebrovascular accident, transient ischemic attack, deep vein thrombosis, pulmonary embolism).

  10.Hereditary or acquired bleeding/thrombotic disorders (e.g., hemophilia, thrombocytopenia).

  11. Urinalysis showing proteinuria ≥++ with 24-hour urine protein >1.0 g. 12. Active infection, unexplained fever ≥38.5°C within 7 days prior to treatment, or baseline leukocyte count >15×10⁹/L.

  13. Congenital or acquired immunodeficiency (e.g., HIV infection). 14. Other factors deemed by the investigator to compromise patient safety or study outcomes (e.g., substance abuse, severe comorbidities, psychiatric disorders, or social circumstances affecting compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
conversion rate | up to 20 weeks
  the conversion rate to curative primary lung lesion resetion in patients with unresectable stage IIIB-IIIC NSCLC following induction chemoimmunotherapy
1-y PFS | within one year
  the proportion of patients without disease progression in one year after the initial dose of chemoimmumotherapy

SECONDARY OUTCOMES:
safety | up to 2 years
  types and incidence of adverse events occurring during the treatment period
the rate of major pathological response (MPR) | up to 20 weeks
  the proportion of patients who achieve MRP among those receiving pneumonectomy
the rate of pathological complete response (pCR) | up to 20 weeks
  the proportion of patients who achieve pCR among those receiving pneumonectomy
PFS | 5 years
  progression-free survival
OS | 5 years
  overall survival
the incidence of radiation pneumonitis | 1-2 years
  the incidence of radiation pneumonitis

OTHER OUTCOMES:
the survival impact of different treatment modalities for contralateral hilar or mediastinal lymph node metastasis | within 5 years
  the survival differences between patients with contralateral hilar or mediastinal lymph node metastasis who received contralateral lymph node radiotherapy versus surgical lymph node dissection

IPD SHARING:
Plan to Share IPD: No